CLINICAL TRIAL: NCT00884780
Title: Development of a New Electronic Measure of Pediatric Pain: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jennifer Verrill Schurman, Co-Director Abdominal Pain Team, Children's Mercy Hospital Kansas City
Other Study IDs: 09 01-020E
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Pediatric Pain
Keywords: Electronic Diary; Body Map; Electronic Measure of Pediatric Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Pain: Children between the ages of 8 and 17 experiencing pain.

SUMMARY:
The purpose of this study is to test the accuracy of a computer-based program to self-report the location and intensity of a child's pain in comparison to a traditional self-report paper and pencil measure and physician physical exam. Using a computer to assess pediatric pain may offer many advantages and improvements in how pediatric pain is diagnosed and treated.

DETAILED DESCRIPTION:
Approximately 1 in 4 children aged 5-18 report experiencing pain. As many as 2 in 3 of these children will develop a significant physical, emotional, social or academic impairment. Recent research has identified pediatric pain as an area where biological, psychological and social treatments can interact to provide substantial changes in pain symptoms. However, there is a lamentable dearth of empirical studies evaluating the efficacy of treatments for chronic pain in children. These findings necessitate more intensive efforts to improve methods on initial assessment and treatment, but an important first step is to improve the sensitivity of outcome evaluation.

Existing measures of pediatric pain have been concerned with symptom intensity and the general locus of pain. Children are traditionally asked to mark with a number or a color the region in which they experience pain. This is helpful for understanding generality that a large area such as the head, joints, or stomach hurts. However, it does not allow the child the option to specify a narrow area of discomfort within a broader region (e.g., upper right quadrant of the stomach). Consequently, current pain instruments may lead to an inaccurate or imprecise understanding of a child's pain, which can adversely impact clinical care of the quality of clinical trials.

The current study will compare a widely used paper-based "pain mapping" tool to a new electronic tool designed by study investigators to capture the same information as the paper measure, while adding more precision regarding pain regions and greater range in terms of pain intensity. We expect that children's responses on these two measures (pencil/paper and electronic) will be generally similar, but we expect that the electronic measure will map more closely onto the Attending Physician's notes regarding discrete pain location, intensity, and/or diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to either APC Clinic or IPM Clinic.
* Child participant is 8-17 years of age.

Exclusion Criteria:

* Child/parent not English speaking.
* Child unable to see computer screen or interact with the keyboard or mouse.
* Parent/child unable or unwilling to provide permission/assent.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Presentation to either Abdominal Pain Clinic or Integrative Pain Management Clinic. A total of ten patients from each clinic, five (5) aged 8-12 and five (5) aged 13-17.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To establish initial acceptability and feasibility of an electronic tool for pain assessment. | One-time standard of care visit.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Friesen, M.D., Study Chair — Children's Mercy Hospital - Gastroenterology:Abdominal Pain Team; Mark Connelly, PhD, Study Chair — The Children's Mercy Hospital: Integrative Pain Medicine Clinic; Joy Weydert, M.D, Study Chair — The Children's Mercy Hospital: Integrative Pain Management Clinic; Jennifer V Schurman, PhD, Principal Investigator — Children's Mercy Hospital Kansas City; Christopher C Cushing, PhD, Study Chair — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States